CLINICAL TRIAL: NCT07301515
Title: Randomised, Double-Blind, Vehicle-Controlled Trial of a Proprietary Daily Antioxidant + SPF Formulation on Mitochondrial DNA Damage in Human Facial Skin
Brief Title: Randomised Controlled Trial of an Antioxidant and Sunscreen Combination Cream for Reducing DNA Damage in Human Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klira Skin (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other); Newcastle-upon-Tyne Hospitals NHS Trust (Other); Skin Analytics Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KLR-MITO-2025-01
Record Dates: First submitted 2025-11-15; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Photoaging; Photodamage; Mitochondrial Damage; Sunscreen; Antioxidants; Preventive Dermatology
Keywords: Photoprotection; Broad-spectrum SPF 50; Encapsulated UV filters; Mitochondrial DNA; Oxidative stress; Facial skin; Vehicle-controlled trial; Randomized double-blind trial; Red algae extract; Resveratrol (bioferment); Vitamin E (tocopherol); Liquorice extract; Skin barrier
MeSH Terms: interventions — Antioxidants

STUDY DESIGN:
Intervention Model Description: Participants are randomized in a parallel assignment to receive either an encapsulated SPF 50 plus multi-antioxidant cream (active) or a vehicle-only cream (comparator). A small, non-randomized observational group continues their usual skincare routine and/or sunscreen use to provide contextual background data. Randomization uses computer-generated block sequences with allocation concealment. Both participants and investigators are blinded to treatment assignment for the randomized arms.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study with multiple levels of masking. Participants, care providers, investigators, and outcome assessors are blinded to treatment allocation. Study creams are dispensed in identical, opaque containers labeled only as "Formulation A" or "Formulation B." The randomization code is maintained by an independent administrator who is not involved in participant interaction, data collection, or analysis. Laboratory personnel and statisticians receive only anonymized, coded samples and datasets. Unblinding will occur only after database lock and completion of all primary analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antioxidant + Sunscreen Cream (Experimental): Participants apply a daily facial cream containing encapsulated broad-spectrum UV filters (SPF 50+, PA++++) combined with an antioxidant complex composed of Phytexcell Liquorice extract (Glycyrrhiza glabra), Resveratrol bioferment, and Vitamin E (tocopherol). The cream is applied once daily in the morning to the full face for 12 weeks.
  Interventions: Combination Product: Antioxidant + Sunscreen Cream
- Vehicle-Only Cream (Placebo Comparator): Participants apply an identical-appearing vehicle cream without UV filters, or antioxidants. The product base, texture, and packaging are identical to the active formulation. It is applied once daily in the morning to the full face for 12 weeks.
  Interventions: Combination Product: Placebo cream

INTERVENTIONS:
Combination Product: Antioxidant + Sunscreen Cream — A daily facial cream containing encapsulated broad-spectrum UV filters (SPF 50+, PA++++) combined with an antioxidant complex composed of Phytexcell Liquorice extract (Glycyrrhiza glabra), Resveratrol bioferment, and Vitamin E (tocopherol). The cream is applied once daily in the morning to the full face (approximately 2 mg/cm²) for 12 weeks.
  Other Names: Proprietary Antioxidant + SPF Formulation
  Arms: Antioxidant + Sunscreen Cream
Combination Product: Placebo cream — An identical-appearing vehicle cream without UV filters or antioxidant actives. The base formulation, texture, and packaging are identical to the active product. Applied once daily in the morning to the full face (approximately 2 mg/cm²) for 12 weeks.
  Other Names: Vehicle cream
  Arms: Vehicle-Only Cream

SUMMARY:
This randomized, double-blind, vehicle-controlled clinical trial investigates whether daily use of an encapsulated SPF 50 formulation containing a multi-antioxidant complex provides greater mitochondrial DNA (mtDNA) protection in human facial skin compared with a vehicle-only cream.

Fifty-two healthy adults will be enrolled during the UK spring and randomized 1:1 to receive either the antioxidant-enriched SPF 50 or a matched vehicle (no SPF, no antioxidants). Participants will apply their assigned product once daily to the full face for 12 weeks under ambient ultraviolet (UV) and oxidative exposure.

Non-invasive cheek swabs collected at baseline and week 12 will be analyzed by blinded quantitative polymerase chain reaction (qPCR) to assess mtDNA integrity (ΔCt = Ct_long - Ct_short).

The primary objective is to determine whether the antioxidant-enriched SPF 50 reduces mtDNA damage compared with vehicle. Secondary objectives include comparing the proportion of "responders" showing reduced mtDNA damage (ΔCt < 0) and evaluating within-participant change among habitual daily sunscreen users.

The trial aims to clarify whether adding antioxidants to high-SPF formulations can strengthen daily photoprotection by mitigating residual oxidative stress not fully blocked by UV filters alone.

DETAILED DESCRIPTION:
Chronic sun exposure generates oxidative stress that damages both nuclear and mitochondrial DNA in skin cells, contributing to photoaging. Mitochondrial DNA is particularly susceptible to ultraviolet- and reactive-oxygen-mediated injury. Even high-SPF sunscreens only partially prevent oxidative stress from UVA, visible, and infrared wavelengths. Combining topical antioxidants with UV filters may enhance cellular protection, but direct in-vivo evidence of mitochondrial benefit during daily use remains limited.

This single-center, randomized, double-blind, vehicle-controlled study will evaluate the effect of a multi-antioxidant, encapsulated SPF 50 formulation on facial mitochondrial DNA integrity during twelve weeks of normal daily use. The study will be conducted during the UK spring to minimize environmental variability in ultraviolet intensity, temperature, and humidity. Healthy adults aged eighteen to seventy years with intact facial skin will be eligible regardless of baseline sunscreen habits. Individuals with active facial dermatologic disease, recent laser or peel procedures within three months, recent use of retinoids, antioxidants, or anti-inflammatory agents within four weeks, pregnancy, lactation, acute illness, or planned high-UV travel will be excluded. Participants taking medications known to affect mitochondrial function must be on stable doses for at least three months before and throughout the study.

Participants will be randomized in a one-to-one ratio to receive either an encapsulated SPF 50 plus multi-antioxidant complex or a vehicle-only cream containing no SPF and no antioxidants. A small non-randomized comparator group may continue their existing skincare routine to contextualize background variability. Study products will be visually identical, coded, and packaged in identical containers to maintain blinding of participants, investigators, and laboratory staff. Each participant will apply the assigned product once daily to the entire face at a standardized dose of approximately two milligrams per square centimeter for twelve weeks. Adherence will be encouraged through written instructions and monitored by self-report and returned product weight.

At baseline and week twelve, a defined two-by-two-centimeter cheek area will be sampled using a sterile synthetic-tipped swab. Samples will be labeled with coded identifiers and analyzed by a blinded external laboratory using a validated long- and short-amplicon quantitative polymerase chain reaction assay. The mitochondrial DNA integrity index, calculated as ΔCt = Ct_long - Ct_short, reflects lesion frequency, where a negative change indicates improved integrity.

The primary outcome is the change in ΔCt from baseline to week twelve between treatment arms. Secondary outcomes include the proportion of participants with ΔCt < 0, the within-participant change among habitual daily sunscreen users compared with their prior routine, and overall safety and tolerability of both products. Efficacy analyses will include all randomized participants with valid paired baseline and week-twelve data. Between-group comparisons will be performed using two-sided parametric and non-parametric tests, and responder proportions will be compared using Fisher's exact test at a significance level of 0.05.

This study will determine whether daily application of an encapsulated SPF 50 formulation containing multiple antioxidants provides superior mitochondrial protection in facial skin compared with vehicle alone, thereby supporting the concept that antioxidant-enriched sunscreens can enhance photoprotection and reduce oxidative stress encountered in everyday life.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-80 years
* Healthy facial skin with no active dermatologic disease
* Willing to apply the assigned product daily for 12 weeks
* Willing to avoid additional facial skincare products during the study period
* Able to attend baseline and week-12 visits for cheek-swab collection
* Willing to maintain stable medication and supplement use throughout the study
* Provided written informed consent

Exclusion Criteria:

* Active facial dermatologic disease or visible facial skin lesions
* Laser, peel, or energy-based facial treatment within the past 3 months
* Use of topical/systemic retinoids, antioxidants, or anti-inflammatory agents within 4 weeks of baseline
* Pregnancy or breastfeeding
* Recent acute illness or infection
* Planned travel to high-UV or sunny destinations during the study period
* Current smoker or regular e-cigarette user
* Participation in another clinical trial within the previous 30 days
* Known allergy or sensitivity to study-product ingredients
* Unstable medical conditions or medications known to affect mitochondrial function (e.g., recent changes in antibiotics, statins, or thyroid medication)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-11-10 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
Difference in Change in Mitochondrial DNA Damage (ΔCt) Between Active and Vehicle Creams Measured by Long-Amplicon Quantitative PCR | Baseline to Week 12
  Mitochondrial DNA (mtDNA) integrity will be assessed from non-invasive cheek swabs using long-amplicon quantitative polymerase chain reaction (qPCR). Two mtDNA fragments are amplified: a long fragment (damage-sensitive) and a short fragment (control for total DNA). ΔCt ("delta-Ct") = Ct_long - Ct_short, where higher values indicate greater mtDNA damage. For each participant, the change in ΔCt from baseline to Week 12 will be calculated. The primary outcome is the between-group difference in this change (Active minus Vehicle), adjusted for baseline values. Negative values denote reduced mtDNA damage with the antioxidant + SPF formulation. Laboratory staff and statisticians are blinded to allocation.

SECONDARY OUTCOMES:
Proportion of Participants With Reduced Mitochondrial DNA Damage (ΔCt < 0) | Baseline to Week 12
  Participants will be classified as "responders" if their change in ΔCt from baseline to Week 12 is < 0, indicating reduced mtDNA damage. The proportion of responders will be compared between randomized arms. Analyses are blinded.
Change in Mitochondrial DNA Damage (ΔCt) From Baseline to Week 12 Among Habitual Daily Sunscreen Users - Active Arm | Baseline to Week 12
  Among participants who reported daily sunscreen use at baseline, change in ΔCt from baseline (reflecting prior sunscreen routine) to Week 12 will be analyzed while using the antioxidant + SPF 50 cream. Negative change denotes less mtDNA damage at Week 12. Paired, blinded analysis.
Change in Mitochondrial DNA Damage (ΔCt) From Baseline to Week 12 Among Habitual Daily Sunscreen Users - Vehicle Arm | Baseline to Week 12
  Among participants who reported daily sunscreen use at baseline, change in ΔCt from baseline (reflecting prior sunscreen routine) to Week 12 will be analyzed while using the vehicle cream without SPF or antioxidants. Positive change denotes greater mtDNA damage at Week 12. Paired, blinded analysis.
Tolerability and Participant-Reported Cosmetic Acceptability | Baseline to Week 12
  Participants will complete structured questionnaires on tolerability (stinging, burning, redness, dryness, breakouts) and cosmetic acceptability (overall appearance, evenness, brightness, texture, and willingness to continue). Change from baseline will be summarized by treatment group. Assessments are blinded to allocation.

CONTACTS AND LOCATIONS:
Overall Officials: Emma Craythorne, Medicine MBChB, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- St John's Institute of Dermatology, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data will be shared, including mtDNA ΔCt values (baseline and week 12), treatment assignment, age, and habitual sunscreen-use category. Questionnaire outcome data and adverse event information will also be available. The shared dataset will exclude all direct identifiers and any genomic sequence data beyond ΔCt metrics.
Supporting Information: SAP, ICF
Time Frame: Available within 12 months after primary completion and for 36 months thereafter.
Access Criteria: Access will be granted upon reasonable written request accompanied by a brief proposal and analysis plan. Requests will be reviewed by the study steering team, and ethics approval or exemption may be required depending on local regulations.